CLINICAL TRIAL: NCT00147927
Title: Using Tailored Emails to Motivate Healthy Behavior, Improve Health Status, & Reduce Health Care Costs in Employee Populations: A Randomized Trial
Brief Title: Using Tailored Emails to Motivate Healthy Behavior Among Employees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Wood Johnson Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 49924
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2007-08-01 (Estimated); Status verified 2007-07

CONDITIONS: Health Behavior
Keywords: email; internet; health promotion; behavior change; health status; work productivity; healthcare cost; employee
MeSH Terms: conditions — Health Behavior

INTERVENTIONS:
Behavioral: Sequential emails and web support

SUMMARY:
The purpose of this research is to evaluate the efficacy of a multi-component email health promotion program on employee adoption of health promoting behaviors and secondarily on health status, work productivity and health care costs.

DETAILED DESCRIPTION:
The Specific Aims are:

* To demonstrate the feasibility and assess the acceptability of email health promotion among diverse employee groups;
* To evaluate short and intermediate-term changes in health behaviors (e.g., daily fruit/vegetable intake, weekly physical activity) at 6 and 12 months;
* To assess change in health status (SF-12), work productivity, and healthcare costs among email program users and controls;
* To identify person predictors of sustained voluntary participation in a 6 month email health promotion program among the workforce population;
* To disseminate the results to maximize influence on e-health promotion, employer health promotion programs, health insurance policy, and research.

ELIGIBILITY:
Inclusion Criteria:

* Adult employee of participating worksite
* Access to desktop computer

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000
Dates: Start 2003-12; Study Completion 2005-12

PRIMARY OUTCOMES:
Physical Activity
Fruit and Vegetable intake

SECONDARY OUTCOMES:
Antecedents to behavior change
Health status
Work productivity
Costs

CONTACTS AND LOCATIONS:
Overall Officials: Patricia D Franklin, MD MPH MBA, Principal Investigator — University of Massachusetts, Worcester

REFERENCES:
- [Background] Daviglus ML, Liu K, Yan LL, Pirzada A, Manheim L, Manning W, Garside DB, Wang R, Dyer AR, Greenland P, Stamler J. Relation of body mass index in young adulthood and middle age to Medicare expenditures in older age. JAMA. 2004 Dec 8;292(22):2743-9. doi: 10.1001/jama.292.22.2743. PMID 15585734
- [Background] Pelletier KR. A review and analysis of the clinical- and cost-effectiveness studies of comprehensive health promotion and disease management programs at the worksite: 1998-2000 update. Am J Health Promot. 2001 Nov-Dec;16(2):107-16. doi: 10.4278/0890-1171-16.2.107. PMID 11727590
- [Background] Aldana SG, Merrill RM, Price K, Hardy A, Hager R. Financial impact of a comprehensive multisite workplace health promotion program. Prev Med. 2005 Feb;40(2):131-7. doi: 10.1016/j.ypmed.2004.05.008. PMID 15533521
- [Background] Glasgow RE, McCaul KD, Fisher KJ. Participation in worksite health promotion: a critique of the literature and recommendations for future practice. Health Educ Q. 1993 Fall;20(3):391-408. doi: 10.1177/109019819302000309. PMID 8307762
- [Background] Lewis RJ, Huebner WW, Yarborough CM 3rd. Characteristics of participants and nonparticipants in worksite health promotion. Am J Health Promot. 1996 Nov-Dec;11(2):99-106. doi: 10.4278/0890-1171-11.2.99. PMID 10163602
- [Background] Grosch JW, Alterman T, Petersen MR, Murphy LR. Worksite health promotion programs in the U.S.: factors associated with availability and participation. Am J Health Promot. 1998 Sep-Oct;13(1):36-45. doi: 10.4278/0890-1171-13.1.36. PMID 10186933
- [Background] Crump CE, Earp JA, Kozma CM, Hertz-Picciotto I. Effect of organization-level variables on differential employee participation in 10 federal worksite health promotion programs. Health Educ Q. 1996 May;23(2):204-23. doi: 10.1177/109019819602300206. PMID 8744873
- [Background] Abrams DB, Boutwell WB, Grizzle J, Heimendinger J, Sorensen G, Varnes J. Cancer control at the workplace: the Working Well Trial. Prev Med. 1994 Jan;23(1):15-27. doi: 10.1006/pmed.1994.1003. PMID 8016028
- [Background] Bureau of Economic Analysis, 2003; Centers for Medicare and Medicaid Services, 2003(b).
- [Background] Roizen MF, Stephenson M. Real Age: Are you as Young as you Can Be? Cliff Street Books 1996.